CLINICAL TRIAL: NCT04175184
Title: The Effects of the Inclusion of Mobilisation With Movement to an Exercise Programme in Patients With Rotator Cuff Related Pain.
Brief Title: Inclusion of Mobilisation With Movement to an Exercise Programme in Rotator Cuff Related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rafael Baeske, Principal investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10534119.5.0000.5345
Record Dates: First submitted 2019-11-15; First posted 2019-11-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain
Keywords: rotator cuff pain; mobilisation with movement; exercises
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Motor Activity | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, placebo-controlled, with a parallel group design
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of participants: participants will be unaware about the specificities of the group allocation. The inclusion of a sham mobilisation with movement (MWM) procedure has the aim to mask the manual therapy procedure. For a naive participant, it is unlikely that he/she might be able to discern the real MWM from the sham MWM. In addition, participants will be requested to avoid discussing the interventions received with the outcome assessor.
  A scale ranging from "treatment under investigation" to "I don´t know" will be used to assess blinding of participants.
  Blinding of outcome assessor: this research assistant will only be responsible for conducting the outcome assessments. He/she will be unaware of group allocation and will also be requested not to discuss any specifics about the treatment programmes with the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. Exercise programme: 2-3 sets of 10-15 repetitions of shoulder girdle and glenohumeral strengthening exercises performed in different positions in addition to three stretching exercises.
  2. Mobilisation with movement (MWM): the participant and physiotherapist will decide one movement more functionally relevant to the patient. Afterwards, attempts of MWM will be applied to different joints in order to identify one particular MWM that improves significantly the movement previously selected. Then, one set of six to ten repetitions will be applied. This process of pragmatically using MWM will be conducted in every session, but from the second session onwards, two to three sets of ten repetitions will be applied, with an interval of sixty seconds between sets. In case of failure to identify an MWM that improves the movement significantly, the patient decides which one seemed to be best and one set of six repetitions will be applied to the onset of discomfort.
  Interventions: Other: Mobilisation with Movement
- Placebo group (Sham Comparator): 1. The exercise programme is exactly the same as the experimental group.
  2. Sham MWM: the participant and physiotherapist will decide together one movement that is more functionally relevant to the patient. Afterwards, a sham MWM (Delgado-Gil et al 2015) will be applied and the movement previously selected will be repeated six times in the first consultation. The participant will be informed that he/she should move to the onset of symptoms, if they occur.This process will be conducted in every session, but from the second session onwards, two to three sets of 10 repetitions will be applied, with an interval of sixty seconds between sets. In case the sham MWM failed to improve the movement significantly, one set of six repetitions will be applied only.
  Interventions: Other: Sham Mobilisation with Movement

INTERVENTIONS:
Other: Mobilisation with Movement — MWM is a pain-free manual therapy procedure that aims to restore full active pain-free range of motion. It consists of an accessory movement performed by the therapist followed by an active movement executed by the patient. The accessory glide might be produced by the therapist´s hands or by a belt. Minor changes in the amount of force or direction of the glide are common to produce better results.
  The MWM procedures will be used pragmatically in this study. Therefore, several attempts might be needed to produce the outcome desired. In the case of the shoulder, they can be applied to the glenohumeral joint, scapulothoracic joint, acromioclavicular joint, cervical and thoracic spines and the rib cage. The decision making process in this study will be based on the outcome observed. The procedure that produced the greatest improvement in active pain-free range of motion will be the one used on that occasion.
  Other Names: MWM; Mobilization with movement
  Arms: Experimental group
Other: Sham Mobilisation with Movement — Sham MWM is a comparator procedure used in this research to control for placebo related mechanisms of action. This procedure has already been used in previous research (Delgado-Gil et al 2015). Briefly, the therapist will stand opposite to the affected shoulder, he/she will place the thenar eminence of the anterior hand on the skin in front of the humeral head, while the posterior hand will rest on the scapula. Both hands will just lightly rest on the skin, no accessory glide will be performed to the humeral head. Then, the participant will move his/her shoulder in the direction previously selected. Shall the procedure elicit pain-free full range of motion, the participant will move their shoulder ten times. Otherwise, the movement should be performed up to the onset of symptoms.
  Other Names: sham MWM; sham Mobilization with movement
  Arms: Placebo group

SUMMARY:
Rotator cuff related pain is considered the main source of musculoskeletal shoulder pain that affects function and produces pain on movement. Amongst the existing physiotherapeutic management approaches, exercise therapy has been recognized as the first line approach. The use of manual therapy in the management of this condition has been debated and studies have shown contradictory results. A specific manual therapy approach, mobilisation with movement (MWM), seems promising in this population as it aims to improve pain-free range of motion and includes active engagement of the participant.

DETAILED DESCRIPTION:
Rotator cuff related pain is a term that includes a diversity of shoulder conditions known as: subacromial impingement syndrome, rotator cuff tendinitis/tendinopathy, rotator cuff tear, bursitis. The use of a broader term is useful as the diagnostic accuracy of special orthopaedic tests have been widely criticised and are unable to identify pathognomonic sources of symptoms in people presenting with shoulder pain. Additionally, even though diagnostic imaging is capable of identifying pathology in patients with rotator cuff related pain, studies demonstrate that their correlation with clinical presentation is questionable.

Shoulder pain is one of the most common sources of musculoskeletal pain that might affect up to 20% of the population. Additional important epidemiological data concerning shoulder pain is the fact that approximately 40% of people complaining of shoulder pain will still be symptomatic after six months. Physiotherapy has an important role in the management of rotator cuff related pain and exercise is the main therapeutic approach when considering pain and functional restriction,

Mobilisation with movement (MWM) is one alternative musculoskeletal approach that focuses on improving active pain-free range of motion. This concept of treatment incorporates a passive accessory glide produced by the clinician, followed by an active movement executed by the patient. Different studies have suggested positive effects of MWM in patients complaining of shoulder pain. On the other hand, other studies reported no superior effects when using MWM in their studies. Several methodological aspects might have influenced this discrepancy in results, such as population, dosage and type of MWM utilized, follow-up period and outcome measures. Due to this uncertainty, the current research aims to further explore the inclusion of MWM to an exercise programme in patients with rotator cuff related pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral shoulder pain of atraumatic origin.
* Complaining of shoulder pain for at least six weeks.
* Scoring at least 3 out 10 on a numeric pain rating scale (0- no pain; 10- worst pain imaginable).
* Pain on active shoulder movement
* Pain provoked by at least three of the following tests: Hawkins-Kennedy, Neer, painful arc, resisted external rotation, empty or full can.
* Participants referred by a specialist under the diagnosis of subacromial impingement syndrome, rotator cuff tendinopathy, partial rotator cuff tears, subacromial pain, bursitis.

Exclusion Criteria:

* Shoulder pain following a traumatic event.
* History compatible with complete rotator cuff and biceps rupture.
* Adhesive capsulitis.
* History of dislocation.
* Glenohumeral osteoarthritis.
* Cancer
* Systemic, local or self-immune inflammatory conditions.
* Previous shoulder or neck surgery.
* Familiar pain provoked by neck movements.
* Presence of radicular signs.
* Use of corticosteroids over the past six months.
* Diagnosis of fibromyalgia.
* Participants with clinical depression
* Participants under treatment for her/his shoulder condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain Disability Index (SPADI). | Changes from baseline and study completion (5 weeks) and 4 weeks follow-up.
  SPADI is a self-reported questionnaire that contains thirteen different items. There are two domains: pain (5 items) and functional activity (8 items). Each item ranges from 0 (no pain / no difficulty) to 10 (worst imaginable pain / so difficult that requires help).
Visual Analogue Scale (VAS) for pain. | Changes from baseline and study completion (5 weeks) and 4 weeks follow-up.
  VAS for pain, is a scale that measures pain level. The scale ranges from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Active pain-free range of motion. | Changes from baseline and study completion (5 weeks).
  Active pain-free range of motion will be assessed for flexion, abduction (Kolber et al, 2011), external rotation (Cools et al, 2014) and hand behind back (Satpute et al, 2016). An inclinometer (Baseline, Enterprises Inc) will be used to measure the ranges of motion.
  All measurements will be conducted to the onset of pain.
Pain pressure threshold | Changes from baseline and study completion (5 weeks).
  Measurements will be collected at three different sides: 5 cm distal to the lateral border of the acromion on both sides over the deltoid muscle, and 10 cm distal to the tibiofemoral joint line, over the tibialis anterior muscle on the unaffected side (Paul et al, 2012). A calibrated digital algometer (Wagner instruments, model FPX 25) will be used to assess the pain pressure threshold.
  An interval of 30 seconds will be respected between measurements.
Global rating scale of change (GROC) | Through study completion and 4 weeks follow-up.
  GROC is designed to measure a patient's improvement or deterioration over time as a result of an intervention.The amplitude of this difference is scored on a numerical or visual analogue scale. In this research a 15 point scale will be used (Kamper et al, 2009).
Expectations of physiotherapy | Change at 3 weeks of treatment from baseline
  The scale to be used in this study to assess expectation has been previously used in patients with shoulder disorders (Chester et al, 2018). Participants will answer the following question: "How much do you expect your shoulder problem to change as a result of physiotherapy treatment?. Please circle one box only".
  Possible answers are: Completely recover, Much improve, Slightly improve, No change, Slightly worse, Much worse, Worse than ever.

OTHER OUTCOMES:
Chronic Pain Self-Efficacy Scale | Baseline
  Self-efficacy is considered an important predictor of patients with shoulder pain (Chester et al, 2018). The domains of pain (5 questions) and function (9 questions) of the chronic pain self-efficacy scale will be used in this study (Salvetti & Pimenta, 2005). Values range from 10 to 100, higher values indicate greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faria, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (2):
- Brazil (2):
  - Albrecht - Clínica Integrada de Reabilitação, São Leopoldo, Rio Grande do Sul
  - Faculdades Integradas de Taquara, Taquara, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis JS. Rotator cuff tendinopathy/subacromial impingement syndrome: is it time for a new method of assessment? Br J Sports Med. 2009 Apr;43(4):259-64. doi: 10.1136/bjsm.2008.052183. Epub 2008 Oct 6. PMID 18838403
- [Background] Hegedus EJ, Goode A, Campbell S, Morin A, Tamaddoni M, Moorman CT 3rd, Cook C. Physical examination tests of the shoulder: a systematic review with meta-analysis of individual tests. Br J Sports Med. 2008 Feb;42(2):80-92; discussion 92. doi: 10.1136/bjsm.2007.038406. Epub 2007 Aug 24. PMID 17720798
- [Background] Hegedus EJ, Cook C, Lewis J, Wright A, Park JY. Combining orthopedic special tests to improve diagnosis of shoulder pathology. Phys Ther Sport. 2015 May;16(2):87-92. doi: 10.1016/j.ptsp.2014.08.001. Epub 2014 Aug 10. PMID 25178255
- [Background] Gismervik SO, Drogset JO, Granviken F, Ro M, Leivseth G. Physical examination tests of the shoulder: a systematic review and meta-analysis of diagnostic test performance. BMC Musculoskelet Disord. 2017 Jan 25;18(1):41. doi: 10.1186/s12891-017-1400-0. PMID 28122541
- [Background] Moosmayer S, Tariq R, Stiris MG, Smith HJ. MRI of symptomatic and asymptomatic full-thickness rotator cuff tears. A comparison of findings in 100 subjects. Acta Orthop. 2010 Jun;81(3):361-6. doi: 10.3109/17453674.2010.483993. PMID 20450423
- [Background] Minagawa H, Yamamoto N, Abe H, Fukuda M, Seki N, Kikuchi K, Kijima H, Itoi E. Prevalence of symptomatic and asymptomatic rotator cuff tears in the general population: From mass-screening in one village. J Orthop. 2013 Feb 26;10(1):8-12. doi: 10.1016/j.jor.2013.01.008. eCollection 2013. PMID 24403741
- [Background] Schwartzberg R, Reuss BL, Burkhart BG, Butterfield M, Wu JY, McLean KW. High Prevalence of Superior Labral Tears Diagnosed by MRI in Middle-Aged Patients With Asymptomatic Shoulders. Orthop J Sports Med. 2016 Jan 5;4(1):2325967115623212. doi: 10.1177/2325967115623212. eCollection 2016 Jan. PMID 26779556
- [Background] Kvalvaag E, Anvar M, Karlberg AC, Brox JI, Engebretsen KB, Soberg HL, Juel NG, Bautz-Holter E, Sandvik L, Roe C. Shoulder MRI features with clinical correlations in subacromial pain syndrome: a cross-sectional and prognostic study. BMC Musculoskelet Disord. 2017 Nov 21;18(1):469. doi: 10.1186/s12891-017-1827-3. PMID 29157224
- [Background] Picavet HS, Schouten JS. Musculoskeletal pain in the Netherlands: prevalences, consequences and risk groups, the DMC(3)-study. Pain. 2003 Mar;102(1-2):167-78. doi: 10.1016/s0304-3959(02)00372-x. PMID 12620608
- [Background] Karel YHJM, Verhagen AP, Thoomes-de Graaf M, Duijn E, van den Borne MPJ, Beumer A, Ottenheijm RPG, Dinant GJ, Koes BW, Scholten-Peeters GGM. Development of a Prognostic Model for Patients With Shoulder Complaints in Physical Therapist Practice. Phys Ther. 2017 Jan 1;97(1):72-80. doi: 10.2522/ptj.20150649. PMID 27538898
- [Background] Abdulla SY, Southerst D, Cote P, Shearer HM, Sutton D, Randhawa K, Varatharajan S, Wong JJ, Yu H, Marchand AA, Chrobak K, Woitzik E, Shergill Y, Ferguson B, Stupar M, Nordin M, Jacobs C, Mior S, Carroll LJ, van der Velde G, Taylor-Vaisey A. Is exercise effective for the management of subacromial impingement syndrome and other soft tissue injuries of the shoulder? A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Man Ther. 2015 Oct;20(5):646-56. doi: 10.1016/j.math.2015.03.013. Epub 2015 Apr 1. PMID 25920340
- [Background] Page MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012224. doi: 10.1002/14651858.CD012224. PMID 27283590
- [Background] Steuri R, Sattelmayer M, Elsig S, Kolly C, Tal A, Taeymans J, Hilfiker R. Effectiveness of conservative interventions including exercise, manual therapy and medical management in adults with shoulder impingement: a systematic review and meta-analysis of RCTs. Br J Sports Med. 2017 Sep;51(18):1340-1347. doi: 10.1136/bjsports-2016-096515. Epub 2017 Jun 19. PMID 28630217
- [Background] Delgado-Gil JA, Prado-Robles E, Rodrigues-de-Souza DP, Cleland JA, Fernandez-de-las-Penas C, Alburquerque-Sendin F. Effects of mobilization with movement on pain and range of motion in patients with unilateral shoulder impingement syndrome: a randomized controlled trial. J Manipulative Physiol Ther. 2015 May;38(4):245-52. doi: 10.1016/j.jmpt.2014.12.008. Epub 2015 Apr 30. PMID 25936465
- [Background] Teys P, Bisset L, Vicenzino B. The initial effects of a Mulligan's mobilization with movement technique on range of movement and pressure pain threshold in pain-limited shoulders. Man Ther. 2008 Feb;13(1):37-42. doi: 10.1016/j.math.2006.07.011. Epub 2006 Oct 27. PMID 17070090
- [Background] Satpute KH, Bhandari P, Hall T. Efficacy of Hand Behind Back Mobilization With Movement for Acute Shoulder Pain and Movement Impairment: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2015 Jun;38(5):324-34. doi: 10.1016/j.jmpt.2015.04.003. Epub 2015 Jun 20. PMID 26099206
- [Background] Guimaraes JF, Salvini TF, Siqueira AL Jr, Ribeiro IL, Camargo PR, Alburquerque-Sendin F. Immediate Effects of Mobilization With Movement vs Sham Technique on Range of Motion, Strength, and Function in Patients With Shoulder Impingement Syndrome: Randomized Clinical Trial. J Manipulative Physiol Ther. 2016 Nov-Dec;39(9):605-615. doi: 10.1016/j.jmpt.2016.08.001. Epub 2016 Nov 6. PMID 27829501
- [Background] Lirio Romero C, Torres Lacomba M, Castilla Montoro Y, Prieto Merino D, Pacheco da Costa S, Velasco Marchante MJ, Bodes Pardo G. Mobilization With Movement for Shoulder Dysfunction in Older Adults: A Pilot Trial. J Chiropr Med. 2015 Dec;14(4):249-58. doi: 10.1016/j.jcm.2015.03.001. Epub 2015 Nov 24. PMID 26793036
- [Background] Martins J, Napoles BV, Hoffman CB, Oliveira AS. The Brazilian version of Shoulder Pain and Disability Index: translation, cultural adaptation and reliability. Rev Bras Fisioter. 2010 Nov-Dec;14(6):527-36. English, Portuguese. PMID 21340248
- [Background] Kolber MJ, Vega F, Widmayer K, Cheng MS. The reliability and minimal detectable change of shoulder mobility measurements using a digital inclinometer. Physiother Theory Pract. 2011 Feb;27(2):176-84. doi: 10.3109/09593985.2010.481011. Epub 2010 Aug 8. PMID 20690872
- [Background] Cools AM, De Wilde L, Van Tongel A, Ceyssens C, Ryckewaert R, Cambier DC. Measuring shoulder external and internal rotation strength and range of motion: comprehensive intra-rater and inter-rater reliability study of several testing protocols. J Shoulder Elbow Surg. 2014 Oct;23(10):1454-61. doi: 10.1016/j.jse.2014.01.006. Epub 2014 Apr 13. PMID 24726484
- [Background] Satpute K, Hall T, Kumar S, Deodhar A. A new method of measuring shoulder hand behind back movement: Reliability, values in symptomatic and asymptomatic people, effect of hand dominance, and side-to-side variability. Physiother Theory Pract. 2016 Oct;32(7):520-7. doi: 10.1080/09593985.2016.1222041. Epub 2016 Sep 12. PMID 27618126
- [Background] Paul TM, Soo Hoo J, Chae J, Wilson RD. Central hypersensitivity in patients with subacromial impingement syndrome. Arch Phys Med Rehabil. 2012 Dec;93(12):2206-9. doi: 10.1016/j.apmr.2012.06.026. Epub 2012 Jul 10. PMID 22789774
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Chester R, Jerosch-Herold C, Lewis J, Shepstone L. Psychological factors are associated with the outcome of physiotherapy for people with shoulder pain: a multicentre longitudinal cohort study. Br J Sports Med. 2018 Feb;52(4):269-275. doi: 10.1136/bjsports-2016-096084. Epub 2016 Jul 21. PMID 27445360
- [Background] SALVETTI, M. G.; PIMENTA, C. A. M. Validação da Chronic Pain Self-Efficacy Scale para a Língua Portuguesa. Rev Psiq Clín, v. 32, n. 4, p. 202, 2005
- [Derived] Baeske R, Hall T, Dall'Olmo RR, Silva MF. In people with shoulder pain, mobilisation with movement and exercise improves function and pain more than sham mobilisation with movement and exercise: a randomised trial. J Physiother. 2024 Oct;70(4):288-293. doi: 10.1016/j.jphys.2024.08.009. Epub 2024 Sep 25. PMID 39327172
- [Derived] Baeske R, Hall T, Silva MF. The inclusion of mobilisation with movement to a standard exercise programme for patients with rotator cuff related pain: a randomised, placebo-controlled protocol trial. BMC Musculoskelet Disord. 2020 Nov 12;21(1):744. doi: 10.1186/s12891-020-03765-6. PMID 33183274